CLINICAL TRIAL: NCT06553638
Title: Evaluation of the Prognostic Impact of Decreased Serum beta2 Microglobulin in the First Year of Follow-up of Myeloproliferative Neoplasia
Brief Title: Evaluation of the Prognostic Impact of Decreased Serum beta2 Microglobulin in the First Year of Follow-up of Myeloproliferative Neoplasia (PRODIGE)
Acronym: PRODIGE
Status: Active, not recruiting | Type: Observational
Sponsor: University Hospital, Brest (Other)
Responsible Party: Sponsor
Other Study IDs: 29BRC24.0132 - PRODIGE
Record Dates: First submitted 2024-08-12; First posted 2024-08-14 (Actual); Last update posted 2024-08-14 (Actual); Status verified 2024-04

CONDITIONS: Myeloproliferative Neoplasm
MeSH Terms: conditions — Myeloproliferative Disorders

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — serum, blood DNA.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
50 patients with a diagnosis of MPN will have an assessment of b2microglobuline at diagnosis and after 1 year. b2mic value decrease will be compared to treatment response.

ELIGIBILITY:
Inclusion Criteria:

* MPN patient diagnosed at one of the participating centers
* over 18 yo

Exclusion Criteria:

* Not able to consent

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Patients with a new diagnosis of MPN
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2024-08-12 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
b2mic decrease level between responders and non-responders | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- Chu Brest, Brest, France

IPD SHARING:
Plan to Share IPD: Yes
All collected data that underlie results in a publication
Supporting Information: Study Protocol
Time Frame: Data will be available beginning three years and ending fifteen years following the final study report completion
Access Criteria: Data access requests will be reviewed by the internal committee of Brest UH. Requestors will be required to sign and complete a data access agreement